CLINICAL TRIAL: NCT06712940
Title: Preventing Youth Firearm Violence in New Orleans: A Hospital-Initiated Community Integrated Approach
Brief Title: Supportive Hospital-Based Intervention for Firearm Trauma
Acronym: SHIFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-1631-UMC; U01CE003384-01 (NIH)
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Gun Violence Prevention; Adolescent Behavior
Keywords: Firearm; Violence prevention; Youth
MeSH Terms: conditions — Adolescent Behavior | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): The experimental arm condition consists of motivational interviewing with case management and firearm safety training with a licensed clinical social worker (LCSW). Motivational Interviewing (MI) is a participant-centered yet directive method for enhancing readiness to change. The purpose of MI is to help an individual articulate their own reasons and develop their own plans for making behavioral change. MI respects these values of self-determination and self-efficacy, and emphasizes the participant's right to make decisions about change. The firearm safety training (FST) will be led by the team's LCSW and include a brief demonstration, identification of reasons why the participant may or may not practice safe storage, and develop a plan moving forward. The FST will integrate MI techniques throughout the session.
  Interventions: Behavioral: Motivational Interviewing and Firearm Safety Training, with Case Management
- Treatment as Usual (No Intervention): Patients assigned to the TAU condition will receive standard care for victims of violence at the Trauma Center. All TAU-assigned patients will be screened by psychiatry consult/liaison staff for posttraumatic symptoms, depression, and substance use. Patients with significant symptoms will be offered pharmacotherapy and/or supportive psychotherapy. Patients will also be provided with a list of community resources available for victims of violence, including mental health and social services.
  Patients in TAU will receive the same information sheet (e.g., job training) provided to patients in the MI condition.

INTERVENTIONS:
Behavioral: Motivational Interviewing and Firearm Safety Training, with Case Management — The basic principles of MI as applied to violence risk reduction in victims of gun violence are as follows: Express Empathy, Develop Discrepancy, Roll with Resistance, and Support Self-Determination/Self- Efficacy. MI practitioners offer themselves as a "consultant" while respecting the participant as the real "expert" in their own life. MI also affirms the patient's ability to make changes and communicates trust in the patient's judgments about readiness and plans for change. Motivational interviewing sessions will occur once a month, for six months with a licensed clinical social worker (LCSW).
  The LCSW will additionally provide case management over the course of the six month study, and a one time firearm safety training that covers safe storage methods. At the end of the firearm safety training, the participant will be offered a biometric lock box for free.
  Arms: Intervention Condition

SUMMARY:
This study is a quasi-experimental design, specifically a non-randomized controlled trial (NCT) designed to test the effects of gun violence reduction intervention including MI for youth ages 16-24 years old who present to the Emergency Department or ICU Spirit of Charity Trauma Center (SCTC) at University Medical Centers or another area hospital in New Orleans, Louisiana following a gunshot injury or stab wound. The study will utilize an enrollment strategy that involves alternating, across recruitment days, the assigned study condition. Thus, Day 1 participants would be enrolled into TAU, Day 2 participants would be enrolled in MI-case management condition, Day 3 participants would be enrolled in TAU, etc. This proposed design will minimize any confounds associated with self-selection while possibly increasing enrollment rate.

Research questions include:

1. Will youth allocated to the MI prevention condition have safer firearm related behaviors and beliefs compared to the TAU control condition at 6 months post- enrollment?
2. Will youth allocated to the MI prevention condition have reduced gun violence recidivism compared to the TAU control condition at 18 months post-enrollment.
3. How do youth's social and normative environments influence their gun behaviors and attitudes?

Researchers will compare intervention and TAU arms to see if there are any differences in outcome measures.

Participants will:

1. complete study eligibility assessment, be assigned to one of two conditions depending on the date of assessment, consent, and enroll in the Emergency Department (ED) or inpatient unit of hospital by a study team member,
2. participate in one of two conditions: MI administered by a licensed clinical social worker, or treatment as usual control group (TAU) administered by a study team member (n=170 per condition)
3. complete three surveys (baseline, 3-month, and 6-month) conducted by a study team member
4. 18-month post examination of participant hospital records
5. have the option to complete a 1-1.5 hour interview, 1-3 months after the 6-month survey is completed (n=50)

DETAILED DESCRIPTION:
The long-term goal of this study is to decrease community rates of youth gun violence. The objective is to test the long-term effects of a hospital-initiated intervention and examine how social contexts influence its adoption and sustained effects. This study will be conducted in collaboration with the Spirit of Charity Trauma Center at University Medical Center to implement a hospital-initiated intervention to reduce gun violence amongst older youth.

The multi-faceted intervention includes motivational interviewing and firearm safety training as part of a broader risk reduction effort involving case management. The proposed study, known as the Supportive Hospital-Based Intervention for Firearm Trauma (SHIFT), will employ a mixed methods approach, including a quasi-experimental study, to test the efficacy of the Motivational Interviewing (MI) intervention compared to treatment as usual (TAU) control condition. The hypothesis of this study is that this harm reduction intervention will be more effective in changing firearm-related behaviors and beliefs than the control condition at 3- and 6-months and reducing gun violence at 18-months post-baseline. If successful, the proposed intervention would significantly reduce gun violence and gun violence recidivism amongst youth in our community. The investigators will test our hypothesis via three specific aims:

1. To establish the effects (at 6 months) of a hospital-initiated, community-integrated practice approach on firearm related behaviors and beliefs amongst older youth (16 to 24 years). Our primary working hypothesis is that youth allocated to the MI prevention condition will have safer firearm related behaviors and beliefs compared to the TAU control condition at 6 months post- enrollment.
2. To establish the effects (at 18 months) of hospital-initiated, community-integrated practice- based approach on rates of gun violence amongst older youth (16 to 24 years). Our primary working hypothesis is that youth allocated to the MI prevention condition will have reduced gun violence recidivism compared to the TAU control condition at 18 months post-enrollment. Gun violence constructs to be measured include hospital readmittance for gun violence wounds, arrest records for gun violence, and frequency of carrying or using a gun.
3. To gain in-depth understanding of older youth's (16 to 24 years) social and normative environments that may influence such a practice. Supplementing quantitative findings with a qualitative study of older youth will more fully capture the social contexts supporting or hindering gun violence behavior changes supported by our practice-based approach. Identifying and examining these factors in-depth will contribute to a more nuanced understanding of how to support the long-term durability of approach effects.

ELIGIBILITY:
Inclusion Criteria:

* 16 to 24 years old
* gunshot wound, stab wound, or assault related blunt force trauma injury treated at University Medical Center
* reside in the state of Louisiana
* capacity to provide voluntary informed consent or assent as approved by the Institutional Review Board of Tulane University

Exclusion Criteria:

* not voluntarily agreeing to participate
* not available to participate in study activities in a private room
* age under 16 or over 24
* do not reside in the state of Louisiana
* not acknowledging English as their first language
* being in the judgment of the trauma surgery service as too physically compromised to participate
* intellectual disability as estimated by clinician judgment following mental status examination
* current psychosis as evidenced by structured clinical interview and mental status examination that are administered on as needed basis
* current legal detention status
* injury was a result of intimate partner violence
* does not have the capacity to provide voluntary informed consent or assent as approved by the Institutional Review Board of Tulane University

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Firearm carriage | At time of enrollment
  Frequency of firearm carriage outside of home
Firearm storage | At time of enrollment
  Categorical description of firearm storage (locked and loaded, locked and unloaded, unlocked and loaded, unlocked and unloaded)
Firearm beliefs | At time of enrollment
  Summary scale of firearm beliefs from a modified version of the Gun Beliefs and Behaviors Scale (GBBS). 7-point Likert scale will be used, and summed to create a composite score where a higher score indicates more positive firearm beliefs. The composite score range will be 0 to 21.
Firearm carriage | 3 months post-enrollment
  Frequency of firearm carriage outside of home
Firearm storage | 3-months post enrollment
  Categorical description of firearm storage (locked and loaded, locked and unloaded, unlocked and loaded, unlocked and unloaded)
Firearm beliefs | 3 months post-enrollment
  Summary scale of firearm beliefs from a modified version of the Gun Beliefs and Behaviors Scale (GBBS). 7-point Likert scale will be used, and summed to create a composite score where a higher score indicates more positive firearm beliefs. The composite score range will be 0 to 21.
Firearm carriage | 6 months post-enrollment
  Frequency of firearm carriage outside of home
Firearm storage | 6 months post-enrollment
  Categorical description of firearm storage (locked and loaded, locked and unloaded, unlocked and loaded, unlocked and unloaded)
Firearm beliefs | 6 months post-enrollment
  Summary scale of firearm beliefs from a modified version of the Gun Beliefs and Behaviors Scale (GBBS). 7-point Likert scale will be used, and summed to create a composite score where a higher score indicates more positive firearm beliefs. The composite score range will be 0 to 21.

SECONDARY OUTCOMES:
Arrest records for gun violence | 18 months post study activity completion
  Number of arrests that an individual experiences from time of study activity completion to 18-months post study activity completion
Hospital readmittance for gun violence wounds | 18 months post study activity completion
  Electronic medical record review to assess for firearm related reinjury

CONTACTS AND LOCATIONS:
Overall Officials: Julia M Fleckman, PhD, MPH, Principal Investigator — Tulane University
Locations (1):
- Tulane School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
IRB approval was not obtained to share IPD with other researchers.

REFERENCES:
- [Background] Lundahl BW, Kunz C, Brownell C, Tollefson D, Burke BL. A meta-analysis motivational interviewing: twenty-five years of empirical studies. Research on Social Work Practice. 2010;20(2):137-160.
- [Background] Purtle J, Rich JA, Fein JA, James T, Corbin TJ. Hospital-Based Violence Prevention: Progress and Opportunities. Ann Intern Med. 2015 Nov 3;163(9):715-7. doi: 10.7326/M15-0586. Epub 2015 Aug 25. No abstract available. PMID 26301734
- [Background] Purtle J, Dicker R, Cooper C, Corbin T, Greene MB, Marks A, Creaser D, Topp D, Moreland D. Hospital-based violence intervention programs save lives and money. J Trauma Acute Care Surg. 2013 Aug;75(2):331-3. doi: 10.1097/TA.0b013e318294f518. No abstract available. PMID 23887566
- [Background] Pino EC, Fontin F, James TL, Dugan E. Mechanism of penetrating injury mediates the risk of long-term adverse outcomes for survivors of violent trauma. J Trauma Acute Care Surg. 2022 Mar 1;92(3):511-519. doi: 10.1097/TA.0000000000003364. PMID 34284465
- [Background] Fein JA, Mollen CJ, Greene MB. The assault-injured youth and the emergency medical system: What can we do? Clinical Pediatric Emergency Medicine. 2013;14(1):47-55.
- [Background] Liebschutz J, Schwartz S, Hoyte J, Conoscenti L, Christian AB Sr, Muhammad L, Harper D, James T. A chasm between injury and care: experiences of black male victims of violence. J Trauma. 2010 Dec;69(6):1372-8. doi: 10.1097/TA.0b013e3181e74fcf. PMID 20838259
- [Background] Mathe N, Johnson ST, Wozniak LA, Majumdar SR, Johnson JA. Alternation as a form of allocation for quality improvement studies in primary healthcare settings: the on-off study design. Trials. 2015 Aug 25;16:375. doi: 10.1186/s13063-015-0904-x. PMID 26303892
- [Background] Mikhail JN, Nemeth LS. Trauma Center Based Youth Violence Prevention Programs: An Integrative Review. Trauma Violence Abuse. 2016 Dec;17(5):500-519. doi: 10.1177/1524838015584373. Epub 2015 Jun 29. PMID 26123004
- See also: firearm homicides data — https://www.cdc.gov/nchs/data/nvsr/nvsr70/nvsr70-04-508.pdf